CLINICAL TRIAL: NCT03588559
Title: Assess the Accuracy of Transtek TMB-1591-A-002 Blood Pressure Monitor in Conformance With the ANSI/AAMI ISO 81060-2 Standard
Brief Title: Clinical Trial of Blood Pressure Monitor in Conformance With the ANSI/AAMI ISO 81060-2 Standard
Acronym: CT_1591-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTS International (Other)
Collaborators: Clinimark, LLC (Other); Guangdong Transtek Medical Electronics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TM-BPM-1801; BTS-TM-BPM-1801 (Other: BTSInternational)
Record Dates: First submitted 2018-06-24; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Blood Pressure
Keywords: Monitors, Blood Pressure
MeSH Terms: interventions — Blood Pressure Determination; Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BPM, TMB-1591-A-002 and Reference Device (Experimental): DUT: Transtek Blood Pressure Monitor TMB-1591-A-002 Reference Device: Baumanometer Desk Mercury Sphygmomanometer. Blood Pressure Measurement with the Transtek BPM TMB-1591-A-002 and with reference device.
  Interventions: Diagnostic Test: Blood Pressure Measurement

INTERVENTIONS:
Diagnostic Test: Blood Pressure Measurement — Measurement blood pressure by Transtek BPM TMB-1591-A-002 and reference device.
  Other Names: Transtek TMB-1591-A-002 and reference device, blood pressure

SUMMARY:
The clinical protocol of the trial:

1. Objective of the trial: To assess the accuracy of device.
2. Test methods and procedures: Perform comparation test on seated position by two devices at the same time.
3. DUT: Transtek Blood Pressure Monitor, Model TMB-1591-A-002, with Cuff (sizes, cm) 15-21, 20-26, 25-34, 25-34(L), 32-43, 32-43(L), 40-55.
4. Reference device: Baumanometer Desk Mercury Sphygmomanometer.
5. Study endpoints: Comply with ANSI/AAMI ISO 81060-2:2013 standard.
6. Statistical methodology used: Standard deviation, Mean error.

DETAILED DESCRIPTION:
1. Introduction:

   Automated blood pressure cuff measurement is the standard of care in numerous medical settings today. This study was designed to assess the accuracy of a previously cleared automated blood pressure cuff system using the same arm sequential dual observer auscultation method. The study was conducted in accordance to ANSI/AAMI/ISO 81060-2:2013 Non-invasive sphygmomanometers - Part 2: Clinical investigation of automated measurement type, the Code of Federal Regulations requirements for Non-Significant Risk Device Investigations and as appropriate ISO 14155: Clinical investigation of medical devices for human subjects - Good clinical practice.
2. Purpose of Clinical Investigation:

   The purpose of this study is to provide supporting documentation for non-invasive blood pressure measurement Accuracy claims for the TMB-1591-A-002 Blood Pressure System with Reusable Cuffs on the intended adult and pediatric population.
3. Clinical Investigation Population:

   Following Salus Independent Review Board (IRB) approval, a total of 90 subjects were screened and enrolled into the study and data was collected. Two subjects were withdrawn from the study and the data was not used in the data analysis. These subjects were removed due to difficulty in hearing the reference blood pressure range (systolic and/or diastolic) and the other was removed due an unstable systolic range. A total of 88 healthy subjects, (53 adult / adolescent and 35 pediatric) ages 3-75yr, arm circumference 15-49.5 cm, systolic blood pressures ranges 79-176.5 and diastolic blood pressure ranges of 49-116 were included in the study for analysis. The study was conducted May 30 - June 16, 2017 to perform an accuracy validation on TMB-1591-A-002 Blood Pressure System with FlexiPortTM Reusable Cuffs.
4. Method:

The requirements for the study were to include a minimum of 85 subjects with a minimum of 35 pediatric subjects 3-12 years of age and the remainder over 12 years of age, with at least 30% being male and 30% being female, and an arm circumference range of 15-55cm where at least six subjects were evaluated in each of the seven cuffs. For the data collection, at least 90% of the subjects needed to contribute 3 paired observations allowing the remaining 10% to be 2 paired observations. A minimum of 255 valid paired observations were needed for the analysis.

This study utilized the same arm sequential method (Dual Observer) in which the observers alternated the measurements for the reference sphygmomanometer and the sphygmomanometer-under test. Each paired reading incorporated the average of the reference reading prior to the device under test and after the device under test. (ANSI/AAMI/ISO 81060-2:2013, Section 5.2.4.2).

The TMB-1591-A-002 Blood Pressure System with FlexiPortTM Reusable Cuffs, (sphygmomanometer-under-test) was designed for use on the upper arm of patients with arm circumferences that range from 15-55cm. Seven cuff sizes were included in the investigation requiring that each cuff size have data collection on at least 6 subjects. Two trained observers (auscultators) simultaneously observed (listened to) the Korotkoff sounds at the brachial artery during the automated blood pressure cuff measurement. The 5th Korotkoff (K5) sound was used to identify diastole for the adult/adolescent subjects and the 4th Korotkoff (K4) sound was used for the pediatric subjects.

The reference sphygmomanometer used in this study [Baumanometer Desk Mercury Sphygmomanometer, SN: CT1573] complied with the requirements of ISO 81060-1 (the maximum error was 1 mmHg per NIST traceable calibration verification.

ELIGIBILITY:
Inclusion Criteria: male,female. Exclusion Criteria: below 3 years old.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurement data | 30 minutes
  Systolic Pressure and Diastolic Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Nagulinie Shukla, Study Chair — Clinimark, LLC
Locations (1):
- Clinimark, LLC, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No